CLINICAL TRIAL: NCT04201717
Title: A Multicenter Randomized Clinical Trial Comparing Surgical Site Infection After Intracorporeal Anastomosis and Extracorporeal Anastomosis for Left Colon Cancer (STARS)
Brief Title: Intracorporeal Anastomosis Versus Extracorporeal Anastomosis for Left Colon Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jilin University (Other)
Responsible Party: Principal Investigator, Dong Yang, Assisted Investigator, Jilin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STARS
Record Dates: First submitted 2019-12-12; First posted 2019-12-17 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-04

CONDITIONS: Colon Cancer
Keywords: total laparoscopic; laparoscopic assisted; intracorporeal anastomosis; extracorporeal anastomosis
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The clinical surgeons, outcome assessors, data recorders, and statisticians will all operate independently. Due to the nature of the surgical interventions, the surgeons will not be blinded to treatment allocation. However, the outcomes assessor who assess or analyze the end point will be blinded. The patients will also be blinded to group allocation to reduce the risk of bias. Unblinding will not be performed unless the finalization of the main data analysis or required for patient's safety. After the data analysis, we will have a blinded interpretation of the study results to minimize misleading data interpretation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic assisted left colectomy (extracorporeal anastomosis group) (Active Comparator): All patients underwent laparoscopic dissection according to the left hemicolon cancer resection standard. lymph nodes and blood vessels, are completely trimmed and resected in an en bloc fashion. A small incision is made in the middle of the abdomen to trim the mesentery, remove the specimen, and complete the anastomosis. After completing the anastomosis, the incision will be sutured.
  Interventions: Procedure: laparoscopic assisted left colectomy (extracorporeal anastomosis group)
- total laparoscopic left colectomy (intracorporeal anastomosis group) (Experimental): All patients underwent laparoscopic dissection according to the left hemicolon cancer resection standard. lymph nodes and blood vessels, are completely trimmed and resected in an en bloc fashion. Mesentery resection is performed under laparoscopy, and anastomosis is completed under laparoscopy. A small incision is made to extract the specimen after the anastomosis is completed.
  Interventions: Procedure: total laparoscopic left colectomy (intracorporeal anastomosis group)

INTERVENTIONS:
Procedure: laparoscopic assisted left colectomy (extracorporeal anastomosis group) — For patients in the control group, the surgeon uses wound edge protectors to exteriorize the colon through a small incision in the midline of the abdomen. A ruler and methylene blue solution are employed to mark the area for colon resection. This guarantees a 10-cm margin from the tumor. Guided by these markers, the marginal vessels and mesentery are divided outside the body. The method of anastomosis is at the surgeon's discretion. A side-to-side anastomosis (including antiperistaltic, isoperistaltic, or overlapping anastomosis) is recommended. Side-to-end or end-to-end anastomosis (sewn by hand or by inserting a circular stapler through the anus or proximal colon) is also allowed. After completing the anastomosis, the incision is sutured. An abdominal drainage tube is inserted at the end of the operation.
  Arms: laparoscopic assisted left colectomy (extracorporeal anastomosis group)
Procedure: total laparoscopic left colectomy (intracorporeal anastomosis group) — In the experimental group, the surgeon will use a 10-cm medical suture and methylene blue solution to mark the resection margin. The marginal vessels and mesentery will be divided inside the body. The proximal and distal colons are resected using a 60mm linear laparoscopic stapler. Side-to-side intracorporeal anastomotic techniques like anti-peristaltic, iso-peristaltic, or overlap methods will be applied. Once the anastomosis is completed, the specimen is retrieved. The surgeon can place the specimen in a sterile plastic bag for retrieval. Alternatively, the surgeon can use a disposable incision retraction fixator to protect the wound. An abdominal drainage tube is inserted.
  Arms: total laparoscopic left colectomy (intracorporeal anastomosis group)

SUMMARY:
This study aims to investigate the effects of intracorporeal anastomosis and extracorporeal anastomosis in laparoscopic-assisted radical left hemicolectomy on surgical site infection. Also consider perioperative recovery, safety, and oncology outcomes.

DETAILED DESCRIPTION:
This is a prospective, randomized controlled trial. In this trial, cases in the intracorporeal anastomosis group and the extracorporeal anastomosis group are allocated at a 1:1 ratio among patients undergoing laparoscopic radical left hemicolectomy. The peri-operative recovery data, complications, oncology outcomes, and survival are compared.

ELIGIBILITY:
Inclusion criteria

1. age between 18 and 80 years;
2. histologically or cytologically confirmed left-sided colon cancer (distal transverse colon, left colic flexure, descending colon, or proximal sigmoid colon);
3. clinical stage T1-4a, N0-2, and M0;
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2;
5. suitable for laparoscopic colectomy;
6. no previous systemic chemotherapy or radiotherapy;
7. willing to provide written informed consent and comply with the research procedures.

Exclusion criteria

1. Have a history of malignant colorectal tumor or have metastatic or multiple carcinoma.
2. Patients with intestinal obstruction, intestinal perforation, intestinal bleeding, etc. who need emergency surgery.
3. Patients who need to undergo combined organ resection or robot-assisted colectomy.
4. Patients who are receiving preoperative neoadjuvant therapy.
5. ASA grade ≥ IV and/or ECOG performance status score > 2.
6. Cardiopulmonary dysfunction (NYHA cardiac function classification II-IV), liver dysfunction (MELD score greater than 12), or kidney dysfunction (serum creatinine above the upper limit of normal);
7. Patients with severe psychiatric illness.
8. Pregnant or lactating women.
9. Patients who have a history of taking hormonal drugs.
10. Diabetic patients whose blood sugar cannot be controlled to be within 6.1 - 8.3 mmol/L.
11. Patients with other clinical and laboratory conditions that are considered by researchers as inappropriate for participating in this trial.

Exit criteria

1. Patients with other non-tumor diseases that prevent them from continuing to receive this treatment regimen.
2. Patients who need emergency surgical resection due to intestinal obstruction, intestinal perforation, intestinal bleeding, etc. after being enrolled in the study.
3. Patients with distant metastasis confirmed by intraoperative exploration or postoperative pathology, including liver, pelvic cavity, ovary, peritoneum, distant lymph node metastasis, etc.
4. Patients who need combined organ resection as determined by intraoperative exploration.
5. Patients who request to withdraw from this study cohort for various reasons after being enrolled in the study, or who cannot complete the study plan and follow-up for various reasons.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2029-07-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Quan Wang, doctor, Principal Investigator — The First Hospital of Jilin University
Locations (12):
- China (12):
  - the First Hospital of Jilin University, Changchun, Jilin
  - Beijing Friendship Hospital, Capital Medical University, Beijing
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing
  - Chinese People's Liberation Army General Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Peking University Cancer Hospital, Beijing
  - The Third Hospital of Jilin University (China - Japan Union Hospital of Jilin University), Changchun
  - Daping Hospital of Army Medical University, Chongqing
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - Fudan University Shanghai Cancer Center (Cancer Hospital Affiliated to Fudan University), Shanghai
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University, Shanghai
  - Shengjing Hospital Affiliated to China Medical University, Shenyang

IPD SHARING:
Plan to Share IPD: Yes
If other researchers want to get the individual participant data of this study and have proper reasons, we'll share the data after the study is completed. Researchers can send an email to the Principal Investigator to ask for permission to use the data.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The Study Protocol, SAP (Statistical Analysis Plan), ICF (Informed Consent Form), and analytic code will be made available following the publication of the primary outcomes. The Individual Participant Data (IPD) will be accessible after the publication of all the long-term secondary outcomes.
Access Criteria: Researchers can send an email to the Principal Investigator to apply for the right to use the data.

REFERENCES:
- [Derived] He L, Li M, Zhang JX, Tong WH, Chen Y, Wang Q. Surgical site infection after intracorporeal anastomosis for left-sided colon cancer: study protocol for a non-inferiority multicenter randomized controlled trial (STARS). Trials. 2022 Nov 22;23(1):954. doi: 10.1186/s13063-022-06914-5. PMID 36415000

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laparoscopic Assisted Left Colectomy (Extracorporeal Anastomosis Group) | Total Laparoscopic Left Colectomy (Intracorporeal Anastomosis Group)
Started | 175 | 175
Completed | 159 | 157
Not Completed | 16 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Total Laparoscopic Left Colectomy (Intracorporeal Anastomosis Group) | Laparoscopic Assisted Left Colectomy (Extracorporeal Anastomosis Group) | Total
Number analyzed (Participants) | 157 | 159 | 316
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [55 to 68] | 61 [53 to 69] | 61 [54 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 52 | 97
  Male | 112 | 107 | 219
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 157 | 159 | 316
bmi [Median (Inter-Quartile Range); unit: kg/m^2] | 24.5 [22.1 to 26.5] | 24.8 [22.9 to 27.1] | 24.6 [22.4 to 26.6]

OUTCOME MEASURES:

1. Primary Outcome: The Count of Participants With Surgical Site Infection (SSI)
Description: The primary outcome was the incidence of SSI based on the Definitions of CDC guidelines: superficial incisional, deep incisional, and organ/space infections . Infections involving both organ/space and the incisional site (superficial or deep) were categorized as organ/space infections. Surgeons and nurses assessed the presence of infection daily during hospitalization. After hospital discharge, all patients were followed up until 30 days after surgery at outpatient clinics to check the wound.
Time Frame: one month after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Total Laparoscopic Left Colectomy (Intracorporeal Anastomosis Group) | Laparoscopic Assisted Left Colectomy (Extracorporeal Anastomosis Group)
Number analyzed (Participants) | 157 | 159
Participants | 15 | 20

2. Secondary Outcome: the Blood Loss
Description: It is defined as the blood loss during operation and is measured in milliliters.
Time Frame: one hour after surgery
Measure: Median (Inter-Quartile Range); unit: ml
Arm/Group | Total Laparoscopic Left Colectomy (Intracorporeal Anastomosis Group) | Laparoscopic Assisted Left Colectomy (Extracorporeal Anastomosis Group)
Number analyzed (Participants) | 151 | 154
ml | 50 [10 to 50] | 50 [10 to 50]

3. Secondary Outcome: the Operating Time
Description: It is defined as the period from cutting the skin to suturing the skin or doing enterostomy. It is measured in minutes
Time Frame: one hour after surgery
Reporting Status: Not Posted

4. Secondary Outcome: the Incidence of Complications
Description: It includes fever of unknown origin, bowel obstruction, anastomotic leakage, SSI, other incisional complications, respiratory complications, urinary complications, cardiovascular and cerebrovascular complications, diarrhea, chylous fistula, intraperitoneal hemorrhage, digestive hemorrhage, gastroparesis, and others (including bacteremia, cholecystitis, ion discharge, pancreatitis, and mental and behavioral abnormalities). Complications are graded according to the Clavien-Dindo classification.
Time Frame: one month after surgery
Reporting Status: Not Posted

5. Secondary Outcome: The Rate of Conversion to Open Surgery
Description: It is defined as an abdominal incision larger than that necessary for specimen extraction.
Time Frame: one hour after surgery
Reporting Status: Not Posted

6. Secondary Outcome: Completeness of Specimens
Description: It is evaluated according to the West classification. The resected specimens will be classified into three groups according to the plane of dissection: mesocolic plane, intramesocolic plane, and muscularis propria plane.
Time Frame: one hour after surgery
Reporting Status: Not Posted

7. Secondary Outcome: Number of Lymph Nodes Dissected
Description: The number of lymph nodes in the mesentery will be calculated. Additionally, the metastatic lymph nodes will be counted.
Time Frame: one week after surgery
Reporting Status: Not Posted

8. Secondary Outcome: First Defecation Time
Description: time to first defecate, measured in days.
Time Frame: one week after surgery
Reporting Status: Not Posted

9. Secondary Outcome: the Incision Length
Description: The incision length is measured with an aseptic ruler at the end of the surgery, after the incision is sutured. It is measured in millimeters.
Time Frame: one hour after surgery
Reporting Status: Not Posted

10. Secondary Outcome: Visual Analogue Scale/Score (VAS)
Description: Pain severity was assessed 48 hours after the operation using a ruler about 10 cm long. The ruler is numbered from 0 to 10. 0-3 points indicate no to mild pain. 4-6 points represent moderate pain. 7-10 points stand for severe pain.
Time Frame: 2 days after surgery
Reporting Status: Not Posted

11. Secondary Outcome: 3-year DFS (Disease-free Survival)
Description: DFS was defined as the time from randomization until the discovery of local recurrence, distant metastasis, or death from the tumor.
Time Frame: three years after the operation
Reporting Status: Not Posted

12. Secondary Outcome: 5-year OS (Overall Survival)
Description: OS was defined as the time from randomization to death due to any cause.
Time Frame: five years after the operation
Reporting Status: Not Posted

13. Secondary Outcome: First Time for Fluid Diet
Description: time to start food intake, measured in days
Time Frame: one week after surgery
Reporting Status: Not Posted

14. Secondary Outcome: Postoperative Hospital Stay
Description: The length of hospital stay after surgery.
Time Frame: one month after surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 30 days after operation
Description: Adverse events studied include intraoperative secondary injuries in patients and serious complications and deaths within 30 days after surgery. An adverse event is defined as any adverse experience that occurs in the subject during the study, regardless of whether it's considered associated with total laparoscopic anastomosis. These include: 1) Accidental secondary damage during surgery. 2) Serious complications after surgery (grade III and above).
Arm/Group | Total Laparoscopic Left Colectomy (Intracorporeal Anastomosis Group) | Laparoscopic Assisted Left Colectomy (Extracorporeal Anastomosis Group)
All-Cause Mortality (participants affected / at risk) | 0/157 | 0/159
Serious Adverse Events (participants affected / at risk) | 10/157 | 6/159
Other Adverse Events (participants affected / at risk) | 13/157 | 24/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Laparoscopic Left Colectomy (Intracorporeal Anastomosis Group) (N=157) | Laparoscopic Assisted Left Colectomy (Extracorporeal Anastomosis Group) (N=159)
Clavien-Dindo grade III or higher complications (Surgical and medical procedures) | 10 (10) | 6 (6)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Laparoscopic Left Colectomy (Intracorporeal Anastomosis Group) (N=157) | Laparoscopic Assisted Left Colectomy (Extracorporeal Anastomosis Group) (N=159)
Clavien-Dindo graded I-II complications (Surgical and medical procedures) | 13 (13) | 24 (24)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT04201717/Prot_SAP_001.pdf